CLINICAL TRIAL: NCT00796146
Title: Establish and Characterize an Acute HIV Infection Cohort in a High Risk Population
Status: Recruiting | Type: Observational
Sponsor: SEARCH Research Foundation (Other)
Collaborators: Armed Forces Research Institute of Medical Sciences, Thailand (Other Government); Thai Red Cross AIDS Research Centre (Other); Yale University (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of California, San Francisco (Other); National Institutes of Health (NIH) (NIH); Johns Hopkins University (Other); University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Nittaya Phanuphak, Nittaya Phanuphak, MD, PhD, Institute of HIV Research and Innovation Foundation, Thailand
Other Study IDs: SEARCH010/ RV 254
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Acute HIV Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, PBMC, cerebrospinal fluid, genital secretions, lymph node biopsy, Gut tissue biopsy
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
To describe clinical, immunological, and virological characteristics of persons with acute HIV infection

1. To describe demographics and behavioral risk factors for those identified with acute HIV infection
2. To describe neurocognitive function and neuroimaging findings in acute HIV infection as well as describe immune response, HIV-1 genotypes and sequences in the cerebrospinal fluid.
3. To describe the number and characteristics of sexual contacts
4. To describe the willingness of acute HIV-infected subjects to allow the tracking of their sexual contacts for voluntary HIV counseling and testing (VCT)
5. To describe immune response, HIV-1 genotypes and sequences in the genital compartment
6. To describe T cell depletion in the gut mucosa in acute HIV infection and describe the changes in gut T cell during follow up
7. To archive samples for future investigations including determination of viral evolution, and cell-mediated and humoral immune responses in peripheral blood and mucosal compartments

DETAILED DESCRIPTION:
This study will establish an acute infection cohort which is predominantly non-subtype B. Description of the early events in HIV infection is critical to HIV vaccine development and understanding HIV-1 immunopathogenesis. The ability to establish this cohort and identify individuals with acute HIV-1 infection would provide the basis for future hypothesis-driven proposals.

Subjects will be recruited at the TRCARC. Subjects seeking VCT will be asked to provide contact information. Blood samples, either plasma or whole blood collected on filter paper (dried blood spots, or DBS) will be screened for acute HIV infection by pooled or individual NAT if non-reactive after screening by an EIA capable of detecting both HIV antibody and antigen (4th generation or sensitive EIA). Additionally, 4th generation reactive samples will be screened with a non-IgM sensitive EIA capable of detecting HIV antibody only (less sensitive EIA) within 1-2 days of sample collection. Those who are found to have acute HIV infection will be asked to enroll in the cohort study. These acute HIV-infected participants will be followed prospectively at week 0, day 2, 3, 5, 7, 10 then weeks 2, 4, 8, 12, 16, 20, 24, then every 12 weeks until the end of the study (maximum of 192 weeks of follow up). Subjects will receive blood testing for CD4, HIV RNA, ALT, creatinine and lipids, and urinalysis. Subjects will be asked to complete a questionnaire on HIV risk behavior. Archiving of plasma and PBMC for future immunologic and virologic testing will be performed. Optional study procedures include 1) collection of genital secretions 2) collection of cerebrospinal fluid 3) brain MRI/MRS without gadolinium 4) sampling of gut-associated lymphoid tissue by colon biopsy 5) genetic testing 6) tracking of and offering VCT to sexual contacts of acute HIV-infected subjects. Subjects are encouraged to be hospitalized for the first 3-7 days for post-procedural observation and for ease of follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old
2. Have protocol-defined acute HIV-1 infection (Tested 4th generation HIV EIA negative and NAT positive or tested 4th generation HIV EIA positive, negative by less sensitive EIA and NAT positive)
3. Understand the study and sign informed consent form. Persons who cannot read will have the consent form read to them by a study staff and they can give informed consent by using thumb print.
4. Availability for follow-up for the planned study duration

Exclusion Criteria:

1. Persons who have a history of a medical or psychiatric disorder by investigator's interview and physical examination according to standard practices, that in the judgment of the investigator(s), would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent.
2. Female participants who are pregnant at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population seeking VCT at the TRCAC will be screened. They are comprised of both men and women of different ages, economic stratus and education level: a large portion of whom are at high risk for HIV infection through commercial sex work and MSM.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2009-04 (Actual); Primary Completion 2033-07 (Estimated); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
Number of HIV and non-HIV related clinical events | It will take approximately 72 months to complete the study. The screening and enrollment is 48 months.

SECONDARY OUTCOMES:
demographics and behavioral risk factors for those identified with acute HIV infection | approximately 72 months to complete the study. The screening and enrollment is 48 months
neurocognitive function and neuroimaging findings in acute HIV infection as well as describe immune response, HIV-1 genotypes and sequences in the cerebrospinal fluid | approximately 72 months to complete the study. The screening and enrollment is 48 months
number and characteristics of sexual contacts | approximately 72 months to complete the study. The screening and enrollment is 48 months
the willingness of acute HIV-infected subjects to allow the tracking of their sexual contacts for voluntary HIV counseling and testing (VCT) | approximately 72 months to complete the study. The screening and enrollment is 48 months
immune response, HIV-1 genotypes and sequences in the genital compartment | approximately 72 months to complete the study. The screening and enrollment is 48 months
T cell depletion in the gut mucosa in acute HIV infection and describe the changes in gut T cells during follow up | approximately 72 months to complete the study. The screening and enrollment is 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandhya Vasan, MD, Study Chair — US Military HIV Research Program
Locations (1):
- Institute of HIV Research and Innovation (IHRI), Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Sacdalan C, Austin C, Varma A, Pinyakorn S, Kroon E, Colby DJ, Chan P, Goh O, Pornpaisakul K, Intasan J, Luekasemsuk T, Robb ML, Chomchey N, Phanuphak N, Ananworanich J, Vasan S, Hsu D; SEARCH 010/RV254 study group. Impaired creatinine-based estimated glomerular filtration rate in Thai individuals switching to dolutegravir: illustrating the role of cystatin C testing to aid clinical decision making. AIDS Res Ther. 2025 Feb 7;22(1):15. doi: 10.1186/s12981-025-00712-0. PMID 39920714
- [Derived] Paul R, Cho K, Bolzenius J, Sacdalan C, Ndhlovu LC, Trautmann L, Krebs S, Tipsuk S, Crowell TA, Suttichom D, Colby DJ, Premeaux TA, Phanuphak N, Chan P, Kroon E, Vasan S, Hsu D, Carrico A, Valcour V, Ananworanich J, Robb ML, Ake JA, Sriplienchan S, Spudich S; RV254/SEARCH 010 Study Team. Individual Differences in CD4/CD8 T-Cell Ratio Trajectories and Associated Risk Profiles Modeled From Acute HIV Infection. Psychosom Med. 2022 Oct 1;84(8):976-983. doi: 10.1097/PSY.0000000000001129. Epub 2022 Jul 6. PMID 36162059
- [Derived] Corley MJ, Sacdalan C, Pang APS, Chomchey N, Ratnaratorn N, Valcour V, Kroon E, Cho KS, Belden AC, Colby D, Robb M, Hsu D, Spudich S, Paul R, Vasan S, Ndhlovu LC; SEARCH010/RV254 and SEARCH013/RV304 study groups. Abrupt and altered cell-type specific DNA methylation profiles in blood during acute HIV infection persists despite prompt initiation of ART. PLoS Pathog. 2021 Aug 13;17(8):e1009785. doi: 10.1371/journal.ppat.1009785. eCollection 2021 Aug. PMID 34388205
- [Derived] Muccini C, Pinyakorn S, Sirivichayakul S, Kroon E, Sacdalan C, Crowell TA, Trichavaroj R, Ananworanich J, Vasan S, Phanuphak N, Colby DJ; RV254 Study Group. Brief Report: Prevalence Trend of Transmitted Drug Resistance in a Prospective Cohort of Thai People With Acute HIV Infection. J Acquir Immune Defic Syndr. 2021 Aug 15;87(5):1173-1177. doi: 10.1097/QAI.0000000000002718. PMID 34229330
- [Derived] Tovanabutra S, Sirijatuphat R, Pham PT, Bonar L, Harbolick EA, Bose M, Song H, Chang D, Oropeza C, O'Sullivan AM, Balinang J, Kroon E, Colby DJ, Sacdalan C, Hellmuth J, Chan P, Prueksakaew P, Pinyakorn S, Jagodzinski LL, Sutthichom D, Pattamaswin S, de Souza M, Gramzinski RA, Kim JH, Michael NL, Robb ML, Phanuphak N, Ananworanich J, Valcour V, Kijak GH, Sanders-Buell E, Spudich S; MHRP Viral Sequencing Core; RV254/SEARCH 010 Study Team. Deep Sequencing Reveals Central Nervous System Compartmentalization in Multiple Transmitted/Founder Virus Acute HIV-1 Infection. Cells. 2019 Aug 15;8(8):902. doi: 10.3390/cells8080902. PMID 31443253
- [Derived] Chan P, Dumrongpisutikul N, Subra C, Colby DJ, Kroon E, Fletcher J, Sacdalan C, Phanuphak N, Valcour V, Ananworanich J, Trautmann L, Spudich S. Neurosyphilis During Acute HIV Infection: A CNS Immunologic and Virologic Characterization. J Acquir Immune Defic Syndr. 2019 Oct 1;82(2):e34-e37. doi: 10.1097/QAI.0000000000002114. No abstract available. PMID 31180994
- [Derived] Chintanaphol M, Sacdalan C, Chottanapund S, Pinyakorn S, Buranapraditkun S, Crowell TA, Kroon E, Manasnayakorn S, Chipman JG, Schacker TW, Michael N, Phanuphak N, Spudich SS, Colby DJ, Ananworanich J. Brief Report: Safety and Tolerability of Inguinal Lymph Node Biopsy in Individuals With Acute HIV Infection in Thailand. J Acquir Immune Defic Syndr. 2018 Oct 1;79(2):244-248. doi: 10.1097/QAI.0000000000001780. PMID 30212436
- [Derived] Ananworanich J, Eller LA, Pinyakorn S, Kroon E, Sriplenchan S, Fletcher JL, Suttichom D, Bryant C, Trichavaroj R, Dawson P, Michael N, Phanuphak N, Robb ML. Viral kinetics in untreated versus treated acute HIV infection in prospective cohort studies in Thailand. J Int AIDS Soc. 2017 Jun 26;20(1):21652. doi: 10.7448/IAS.20.1.21652. PMID 28691436
- [Derived] de Souza MS, Pinyakorn S, Akapirat S, Pattanachaiwit S, Fletcher JL, Chomchey N, Kroon ED, Ubolyam S, Michael NL, Robb ML, Phanuphak P, Kim JH, Phanuphak N, Ananworanich J; RV254/SEARCH010 Study Group. Initiation of Antiretroviral Therapy During Acute HIV-1 Infection Leads to a High Rate of Nonreactive HIV Serology. Clin Infect Dis. 2016 Aug 15;63(4):555-61. doi: 10.1093/cid/ciw365. Epub 2016 Jun 17. PMID 27317797